CLINICAL TRIAL: NCT04509544
Title: Patient's Preferences and Satisfaction About Physical Therapy Reported by Individuals With Cerebral Palsy and Families: ESPaCe, a National Survey in France.
Brief Title: Satisfaction and Preferences About Motor Rehabilitation in People With Cerebral Palsy: ESPaCe, a French Survey
Acronym: ESPaCe
Status: Completed | Type: Observational
Sponsor: Fondation Paralysie Cérébrale (Other)
Collaborators: Kappa Santé (Industry); Envoludia (Unknown); FFAIMC (Unknown); CNSA (Unknown); KLESIA (Unknown); Fondation L'Oréal (Unknown); SESEP (Unknown)
Responsible Party: Sponsor
Other Study IDs: ESPaCe
Record Dates: First submitted 2020-07-07; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy (CP)
Keywords: Physiotherapy; Satisfaction; Unmet needs; Motor Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This national cross-sectional ESPaCe survey (Enquête Satisfaction Paralysie Cérébrale) was conducted to evaluate perceived needs, barriers and expectations regarding Motor Rehabilitation services further to a preliminary qualitative work.

From June 2016 to June 2017, participants answered a web-based or postal questionnaire, by themselves or with the help of a family member.

DETAILED DESCRIPTION:
ESPaCe was a cross-sectional national survey designed to collect data on Cerebral Palsy (CP) motor rehabilitation from individuals with CP and their families in France.

Needs, barriers and expectations regarding PT services were identified in a series of standardised individual interviews and group discussions developed by a multidisciplinary group composed of individuals with cerebral palsy, families, professional organisation representatives, therapists and rehabilitation specialists, described as "ESPaCe working group". The issues identified in the preparatory qualitative work were structured in a questionnaire and tested in a feasibility study.This study was carried out in accordance with the Code of Ethics of the World Medical Association (Declaration of Helsinki). Informed consent was not required for this survey according to current French legislation.The study included all individuals with cerebral palsy aged 2 y.o. or more, whether they were receiving physiotherapy (PT) services at the time of the survey or not. CP features were self-reported. Eligibility was confirmed by cross-checking the responses to questionnaire items related to history, diagnosis and clinical description of CP. The questionnaire was completed either by individuals with cerebral palsy, a family member or a caretaker.

Participants were described with the following characteristics: age, gender, Gross Motor Function Classification System (GMFCS) level, CP subtype, associated impairments, frequency of pain, mother education (as a proxy for socio-economic status), and PT service provider.

Participation in the ESPaCe survey was promoted through local and national patient advocacy groups and professional networks. The questionnaire was completed online or mailed-in. Data collection was open from June 2016 to June 2017.Participation in the ESPaCe survey was promoted through local and national patient advocacy groups and professional networks.

ELIGIBILITY:
Inclusion Criteria:

* Anyone living in France with a motor impairment consistent with the definition of Cerebral Palsy (whether undergoing or not motor rehabilitation sessions)

Exclusion Criteria:

* Individuals who were not diagnosed with CP or when descriptive information provided in the survey regarding motor impairment was insufficiently detailed or did not meet the definition of CP (e.g., progressive disorders).
* Individuals for whom a questionnaire was already completed by a family member or caregiver

Of note main analyses will be run for participants > 2 years old (data for participants < 2 y o considered as exploratory data)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals living in France with a motor impairment consistent with the definition of Cerebral Palsy
Sampling Method: Non-Probability Sample
Enrollment: 1159 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Determinants of satisfaction with motor rehabilitation in people with cerebral palsy | Day 1
  Validated French version of Client Satisfaction Questionnaire (CSQ-8)The CSQ-8 includes 8 items, each rated on a 4-point Likert scale, ranging from 1 to 4. The CSQ-8 total score ranges from 8 to 32. A higher score represents greater satisfaction.
Perceived needs, barrier to access and key expectations for physiotherapy services and associated motives | Day 1
  Likert scale ranging from 0 (never/not at all) to 5 (always/very high); Higher scores mean a worse outcome
Physiotherapy practices | Day 1
  Weekly frequency and duration (min) of physiotherapy sessions

SECONDARY OUTCOMES:
Analysis of the content of the free-text responses (ancillary study of ESPaCe) | Day 1
  Participants' comments were coded and compiled into themes using a text-mining approach allowing to provide context to supplement the results from the closed questions as well as identify any issues or opinions that were not covered by the closed questions.

CONTACTS AND LOCATIONS:
Overall Officials: Javier De La Cruz, MD, Study Chair — Health Research Institute Imas12, Madrid, Spain; Maria BODORIA, MD, Study Director — Fondation Paralysie Cérébrale

IPD SHARING:
Plan to Share IPD: No
Satisfaction, perceived unmet needs, barriers and expectations about motor rehabilitation of children, adolescents and adults with cerebral palsy to be provided as a function of age and GMFCS

REFERENCES:
- [Result] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- See also: rigin, foundations, rationale, governance of ESPaCe: A national survey on unmet needs and expectations' prioritization about motor rehabilitation reported by people with cerebral palsy and their family. Motricité cérébrale 2018;39(2):44-52. — https://doi.org/10.1016/j.motcer.2018.03.002
- See also: Determinants of satisfaction with motor rehabilitation in people with cerebral palsy: A national survey in France (ESPaCe) — https://doi.org/10.1016/j.rehab.2019.09.002